CLINICAL TRIAL: NCT02670980
Title: Compensation for Blindness With the Intelligent Retinal Implant System (IRIS V2) in Patients With Retinal Dystrophy
Acronym: IRIS 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Science Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPP1
Record Dates: First submitted 2016-01-04; First posted 2016-02-02 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Retinitis Pigmentosa; Cone Rod Dystrophy; Choroideremia
Keywords: Retina Implant; Visual Prosthesis
MeSH Terms: conditions — Retinitis Pigmentosa; Cone-Rod Dystrophies; Choroideremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Retina Implant (Experimental): Intelligent Retinal Implant System
  Interventions: Device: Intelligent Retinal Implant System

INTERVENTIONS:
Device: Intelligent Retinal Implant System

SUMMARY:
This study evaluates the safety and effectiveness of the Intelligent Retinal Implants System (IRIS V2). Blind patient suffering from Retinitis Pigmentosa, Cone Rod Dystrophy, or Choroideremia are implanted with an Intelligent Retinal Implant Systeme. All subjects undergo ophthalmological examinations in predefined intervals after implantation. Ophthalmological examinations include funduscopy, slit lamp examination and OCT. All adverse events are recorded and analyzed. Efficacy is measured using functional vision and visual function tests before and after implantation as well as with the system on and system off.

ELIGIBILITY:
Inclusion Criteria:

* Is 25 years or older at the date of enrolment
* Has a confirmed diagnosis of retinitis pigmentosa, choroideremia or cone-rod dystrophy
* Has a visual acuity of logMAR 2.3 or worse in both the eyes as determined by a Square Grating scale.
* Has functional ganglion cells and optic nerve activity
* Has a memory of former useful form vision
* Understands and accepts the obligation to present for all schedule follow-up visits.

Exclusion Criteria:

* Has a history of severe glaucoma, uveitis, optic neuropathy or any confirmed damage to the optic nerve and/or visual cortex related to the projected implanted eye,
* Has any disease (other than study allowed diseases) or condition that affects retinal function of the study eye (e.g., central retinal artery/vein occlusion, end-stage diabetic retinopathy, current or prior retinal detachment, infectious or inflammatory retinal disease, etc.),
* Has any disease or condition that prevents adequate visualization of the retina of the study eye including, but not limited to, corneal degeneration that cannot be resolved prior to implantation,
* Has any disease or condition of the anterior segment of the study eye that prevents adequate physical examination (e.g., ocular trauma, etc.),
* Has severe nystagmus,
* Has any ocular condition that leads him or her to eye rubbing,
* Has any disease or condition that precludes the understanding or communication of the informed consent, study requirements or test protocols (e.g., deafness , multiple sclerosis, amyotrophic lateral sclerosis, neuritis, etc),
* Has a history of epileptic seizure,
* Has a history of chronic or recurrent infection or inflammation that would preclude participation in the study,
* Has a known sensitivity to the contact materials of the implant (platinum and parylene),
* Presents with hypotony in the study eye,
* Presents with hypertony in the study eye,
* Is pregnant or lactating,
* Has another active implanted device (e.g. cochlear implant) or any form of metallic implant in the head (other than dental work) that may interfere with the device function,
* Has a diagnosis requiring an active implant (e.g., cardiac pacemaker, vagus nerve implant, etc.),
* Has active cancer or a history of intraocular, optic nerve or brain cancer and metastasis,
* Is an immune-suppressed subject (e.g., due to HIV positive diagnosis, etc.),
* Is carrier of multi-resistant germs,
* Requires the use of any of the following medications:

  * Antimetabolites,
  * Thrombocyte aggregation reducing therapies (10 days prior until 3 days after surgery),
  * Oral anticoagulants (5 days before until 3 days after surgery),
* Is participating in another investigational drug or device study,
* Has any health concern that makes general anaesthesia inadvisable; Patients with an ASA-Score (or equivalent) of 3 or higher are excluded from the study,
* Is likely requiring MRI scans subsequent to implantation and prior to explantation,
* Is likely requiring therapeutic ultrasound subsequent to implantation and prior to explantation of the Retinal Implant.
* Patients with recurrent or chronic inflammations or infections are excluded from the study. Specifically patients with the following disorders are excluded:

  * Common inflammation - severe chronic and consuming diseases that frequently associated with infection (e.g. Crohn disease, Whipple's disease)
  * Chronic inflammation of the skin in the area of the eye (e.g. dermatitis, rosacea, infection of the skin, herpes zoster)
  * Chronic inflammation in the area of the eye (e.g. herpes of cornea and/or conjunctiva, recurrent blepharoconjunctivitis, hordeolum, chalazion)
* Has a severe psychological disorder. When in any doubt, an expert assessment needs to be arranged to clarify whether the patient's psychological health is suitable for the trial.
* Has severe renal, cardiac, hepatic etc. organ diseases.
* Has eye AP dimension that are incompatible (less than 20.5 or larger than 25mm) with the implant or head dimension that are incompatible with the Visual Interface. Please make sure that the size of the eye socket allows an implantation of the extra ocular part which has a thickness of 5mm.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events according to ISO14155 | up to 36 month
  All subjects undergo ophthalmological examinations in predefined intervals after implantation. Adverse event are rated to be serious or non-serious according ISO14155

SECONDARY OUTCOMES:
Visual acuity | up to 36 month
  Measure probable benefit with square wave grating test
Square localization | up to 36 month
  Measure probable by measuring the error in localizing a white square on black background.
Functional Vision | up to 36 month
  Measure probable benefit e.g. by Functional Picture Assessment. The number of errors subjects make in detecting objects or persons on standardized pictures is measures. Other test may be developed during the study.

CONTACTS AND LOCATIONS:
Locations (9):
- Medical University of Graz, Graz, Austria
- France (3):
  - Clinique Ophtalmologique du CHU de Nantes, Nantes
  - CHU Nimes, Service Ophtalmologie (France)/ Hopital Gui de Chauliac, CHU Montpelier, (France), Nîmes
  - Hopital des Quinze Vingts/Fondation Ophtalmologique A. De Rothschild, Paris
- Germany (3):
  - Dept. of Ophthalmology, University of Bonn, Bonn
  - Universitäts KlinikumKlinik für Augenheilkunde Freiburg, Freiburg im Breisgau
  - Klinik und Poliklinik für Augenheilkunde Hamburg -Eppendorf, Hamburg
- Instituto de Microcirugia Ocular, Barcelona, Spain
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No